CLINICAL TRIAL: NCT06209762
Title: Investigation of the Effects of Inspiratory Muscle Training in Addition to Core Stabilization Exercises on Core Endurance, Functional Capacity, Pain Intensity, Disability, Quality of Life and Sleep Quality in Patients With Mechanical Low Back Pain.
Brief Title: Investigation of the Effects of Inspiratory Muscle Training on Patients With Mechanical Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GulceB
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Mechanical Low Back Pain
Keywords: Mechanical Low Back Pain; Inspiratuar Muscle Training; Core Stabilization Exercise
MeSH Terms: conditions — Low Back Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator)
  Interventions: Other: Exercise
- Inspiratuar Muscle Education Group (Experimental): Patients in this group will have 10 repetitions of slow diaphragmatic deep breathing exercises followed by core stabilization exercises. Then, IMT will be applied with a respiratory muscle training device. In this training, the difficulty of the exercise will be increased by starting from 40% of the MIP value measured during the evaluation and following the values of 60% and 80% according to tolerance. In addition to physical therapy sessions three days a week for eight weeks, patients will be asked to do this exercise five days a week in the morning and evening.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The core stabilization exercise program, which is individually prescribed and structured, will be applied for 8 weeks. The level of exercises will be increased over time according to the patient's condition. Exercises will be taught to patients. It will be carried out under the supervision of a physiotherapist three days a week for 8 weeks. On the remaining days, the patient will be asked to do it himself.

SUMMARY:
There are many conservative treatment methods for the treatment of mechanical low back pain and they continue to be developed. The aim of this study is to examine the effects of inspiratory muscle training, which can be added to these treatment methods, on muscle endurance, functional capacity, pain intensity, disability, quality of life and sleep quality in people with mechanical low back pain.

DETAILED DESCRIPTION:
When initial assessment will be completed, patients will be assigned to one of two possible sequences by simple randomization: study group (SG) or control group (CG).

All participants will receive the core stabilization exercise program designed for mechanical low back pain for 8 weeks. Additionally, the study group will receive inspiratory muscle training for 8 weeks.

All studies will be evaluated both at the beginning and end of the study in terms of pain, quality of life, sleep quality, disability level, muscle endurance and functional capacity. All data will be collected by the same physiotherapist at baseline and at the end of the study (8 weeks). The same physiotherapist will also supervise the exercises and inspiratory training.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18-65
* Applying to the physical therapy unit with the diagnosis of mechanical low back pain (Lumbal disc herniation, spinal stenosis, spondylolisthesis, facet joint pain, discogenic pain, sacroiliac joint pain, myofascial pain, lumbar osteoarthrosis)
* Ability to adapt to exercise commands and understand assessment questions
* Volunteering to participate in research

Exclusion Criteria:

* Those with cooperation and communication problems
* Complaining of acute or chronic musculoskeletal pain other than low back pain
* Having a chronic disease (hypertension, diabetes, chronic obstructive pulmonary disease (COPD), previous cerebrovascular accident (CVO), heart, neurological and rheumatological problems)
* Sequestrated and extruded hernia
* Receiving physical therapy in the last 2 months
* Having a history of recent surgery (spine, abdomen, upper and lower extremity surgeries)
* Being obese (Body mass index ≥30 kg/m2)
* Contagious and vascular diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-12-26 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 8 weeks
  Pain intensity will be measured with this scale.
Oswestry Disability Index | 8 weeks
  Disability level will be measured with this scale
Maximum Inspiratuar Pressure | 8 weeks
  It will be used to evaluate participants' inspiratory muscle strength.
Core Activation | 8 weeks
  It will be used to evaluate the participants' core muscle strength.
2 Minute Walking Test | 8 weeks
  It will be used to evaluate the functional capacity of participants.
Pittsburgh Sleep Quality Index | 8 weeks
  It will be used to evaluate participants' sleep quality.
Short-Form 12 | 8 weeks
  It will be used to evaluate participants' quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University, Ataşehir, Istanbul, Turkey (Türkiye)